CLINICAL TRIAL: NCT06809517
Title: A Phase I/II Clinical Study of Intrathecal Combination Therapy With the PD-1/VEGF Bispecific Antibody and Pemetrexed for Leptomeningeal Metastasis
Brief Title: Intrathecal PD-1/VEGF Bispecific Antibody Plus Pemetrexed for Leptomeningeal Metastasis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Pan, Professor, Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IT-P-AK112
Record Dates: First submitted 2025-01-26; First posted 2025-02-05 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-01

CONDITIONS: Leptomeningeal Metastasis; Intrathecal Drug Delivery
Keywords: Leptomeningeal metastasis; PD-1/VEGF Bispecific Antibody; Pemetrexed
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intrathecal PD-1/VEGF Bispecific Antibody plus Pemetrexed (Experimental): This study is a prospective, single-arm, Phase I/II clinical trial. The primary objective is to determine the recommended Phase II dose (RP2D) for the intrathecal combination of PD-1/VEGF bispecific antibody with pemetrexed and and safety based on the incidence of treatment-related adverse events. Clinical response rate (CRR), progression-free survival related to leptomeningeal metastasis (LMPFS) and overall survival (OS) are also evaluated. Patients will have cerebrospinal fluid (CSF) and blood specimen collection for the evaluation of predictors (clinical, molecular, and/or immune) of the efficacy and safety of this regimen.
  Interventions: Drug: AK112; Drug: Pemetrexed (Alimta)

INTERVENTIONS:
Drug: AK112 — Intrathecal injection of PD-1/VEGF bispecific antibody was administered every two weeks for six weeks during the induction phase, followed by monthly injections during the maintenance phase, until recurrence or death.
Drug: Pemetrexed (Alimta) — Pemetrexed was administrated by intrathecal injection, first as induction therapy, twice per week for 2 weeks, followed by consolidation therapy, once per week for 4 weeks, then maintenance therapy, once per month until the patient's death, leptomeningeal metastasis progresses, or intolerable severe adverse events occurred.

SUMMARY:
Leptomeningeal metastasis, characterized by tumor cells infiltrating and proliferating in the subarachnoid space, represents a distinct pattern of central nervous system involvement and is a fatal complication of malignant tumors.

This phase I/II study is to evaluate the recommended dose, safety, feasibility, and therapeutic response of intrathecal PD-1/VEGF bispecific antibody plus pemetrexed in patients with leptomeningeal metastasis.

DETAILED DESCRIPTION:
Leptomeningeal metastasis represents a severe complication of advanced malignancies, for which intrathecal chemotherapy remains the mainstay treatment. The preliminary results from our previous study on PD-1 combined with pemetrexed intrathecal administration showed safety and feasibility for leptomeningeal metastasis from solid tumors with potential activity. In recent years, targeted therapy and immunotherapy has been widely used for the treatment of solid tumors. As the world's first PD-1/VEGF bispecific antibody, ivonescimab ((AK112) has shown superior systemic efficacy compared to conventional VEGF targeted therapy combined with immunotherapy, while maintaining a favorable safety profile. The primary objectives are to determine the recommended dose of intrathecal ivonescimab in combination with pemetrexed and to assess safety based on the incidence of treatment-related adverse events. Clinical response rate, progression-free survival related to leptomeningeal metastasis, and overall survival are also evaluated. Patients undergo cerebrospinal fluid and blood specimen collection to evaluate potential clinical, molecular, and/or immune predictors of treatment efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of solid tumors;Cerebrospinal fluid cytopathology is positive.
2. Male or female aged between 21 and 75 years; Normal liver and kidney function; WBC≥4000/mm3, Plt≥100000/mm3.
3. No history of severe nervous system disease; No severe dyscrasia.

Exclusion Criteria:

1. Any evidence of nervous system failure, including severe encephalopathy, grade 3 or 4 leukoencephalopathy on imaging, and Glasgow Coma Score less than 11.
2. Any evidence of extensive and lethal progressive systemic diseases without effective treatment.
3. Obvious bleeding tendency; Patients with hemorrhage (NCI-CTCAE v5.0 greater than grade 2), coagulation disorder, hypertensive crisis, and severe arterial thrombosis.
4. A history of HIV or AIDS, acute or chronic hepatitis B or C infection, previous anti-PD1 therapy-induced pneumonitis, or have ongoing >Grade 2 adverse events of such therapy; or ongoing autoimmune disease that required systemic treatment in the past 2 years.
5. The first month to treatment, as well as during induction and consolidation therapy, new drugs effective against leptomeningeal metastases were used, excluding those previously administered. These primarily included small molecule targeted therapies, such as EGFR-TKI/ALK-TKI drugs like Osimertinib and Lorlatinib.
6. Patients with poor compliance or other reasons that were unsuitable for this study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
PR2D | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  The recommended phase II dose. The dose limiting toxicity was defined as ≥ grade 3 neurological toxicities (e.g., chemical meningitis) or other grade 4 toxicity.
Incidence of treatment-related adverse events | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The incidence of treatment-related adverse events were measured for determining tolerability and safety. Adverse events (AEs) are evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE). Events of grade 3-5 are defined as moderate and severe adverse events.

OTHER OUTCOMES:
Clinical response rate | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  The response assessment in neuro-oncology criteria (RANO) proposal for response criteria of leptomeningeal metastasis was used to assess the clinical response in this study.
Progression-free survival related to leptomeningeal metastasis (LMPFS) | From date of treatment until the date of first documented leptomeningeal metastasis progression or date of death from any cause, whichever came first, assessed up to 6 months
  LMPFS was defined as time from the start of treatment until leptomeningeal metastasis progression or death. The leptomeningeal metastasis progression was determined based on the RANO proposal evaluation criteria which have been established and published on Neuro Oncol.
Overall survival(OS) | From the enrollment of this study until date of death from any cause, whichever came first, or the last follow-up，assessed up to 6 months.
  Overall survival was recorded since the date of patient enrollment. All patients were followed up until death or the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Pan, PhD,MD, Principal Investigator — The Affiliated HuizhouHospital, Guangzhou Medical University
Locations (1):
- The Affiliated Huizhou Hospital, Guangzhou Medical University, Huizhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No